CLINICAL TRIAL: NCT04881552
Title: Incidence, Clinical Characteristics and Prognosis of Patients With ST-segment Elevation Myocardial Infarction (STEMI) and Spontaneous Coronary Reperfusion in the Modern Antithrombotic Strategy Area
Acronym: STEMI
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0232
Record Dates: First submitted 2021-05-05; First posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Coronary Syndrome
MeSH Terms: conditions — Angina, Unstable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: non-spontaneous reperfusion group at initial emergency coronary angiography (TIMI flow grade 0-II)
- Arm 2: spontaneous reperfusion group at initial emergency coronary angiography (TIMI flow grade III)

SUMMARY:
The rapid and complete restoration of coronary flow is a key issue in the management of STEMI. Primary percutaneous coronary intervention (PCI) is the preferred reperfusion strategy associated with antithrombotic drugs.

In daily practice, it is not rare that some patients may achieve reopening of the culprit artery without undergoing any mechanical reperfusion therapy, which is called " spontaneous reperfusion ". The latter is associated with improved outcomes in several studies but none of these studies were done in the modern antithrombotic strategy area including new P2Y12 inhibitors. The aim of this study is to report the incidence, characteristics and outcomes of consecutive patients with STEMI admitted for coronary angiography with angiographic clinical evidence of spontaneous reperfusion in the modern medical antithrombotic strategy associated with primary PCI.

ELIGIBILITY:
Inclusion criteria:

* Older than 18 years old.
* patients with ongoing (within 12 hours after onset of symptoms) STEMI admitted for coronary angiography and receiving preloading dose of aspirin, heparin and P2Y12 inhibitor

Exclusion criteria:

* Patients with thrombolysis treatment before angiography
* Patients with cardiac arrest without ST-segment elevation on ECG after resuscitation
* Patients with myocardial infarction outside of acute phase (pain lasting more 12 hours)
* Patients with mental disease
* Patients not living in France

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with ongoing (within 12 hours after onset of symptoms) STEMI admitted for coronary angiography and receiving preloading dose of aspirin, heparin and P2Y12 inhibitor
Sampling Method: Non-Probability Sample
Enrollment: 302 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Incidence of initial spontaneous coronary TIMI flow grade III | At admission
  Incidence of initial spontaneous coronary TIMI flow grade III on coronary angiography before PCI in patients admitted for STEMI during a 6 month study period

SECONDARY OUTCOMES:
Biological parameters | at 6 months
  biological parameters in the 2 groups of patients with or without spontaneous reperfusion including troponin pic at admission and during hospitalization stay Type and delay of administration of the antithrombotic preloading therapy in the 2 groups Clinical follow -up regarding major cardiovascular events at 6 months follow-up in the 2 groups
Biological parameters | at 12 months
  biological parameters in the 2 groups of patients with or without spontaneous reperfusion including troponin pic at admission and during hospitalization stay Type and delay of administration of the antithrombotic preloading therapy in the 2 groups Clinical follow -up regarding major cardiovascular events at 12 months follow-up in the 2 groups
Clinical events | at 6 months
  Clinical events in the 2 groups of patients with or without spontaneous reperfusion including troponin pic at admission and during hospitalization stay Type and delay of administration of the antithrombotic preloading therapy in the 2 groups Clinical follow -up regarding major cardiovascular events at 6 months follow-up in the 2 groups
Clinical events | at 12 months
  Clinical events in the 2 groups of patients with or without spontaneous reperfusion including troponin pic at admission and during hospitalization stay Type and delay of administration of the antithrombotic preloading therapy in the 2 groups Clinical follow -up regarding major cardiovascular events at 12 months follow-up in the 2 groups

CONTACTS AND LOCATIONS:
Overall Officials: Florence Leclercq, PU PH, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC